CLINICAL TRIAL: NCT05537441
Title: Precision Vaccine Promotion in Underserved Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of California, Los Angeles (Other); Los Angeles County Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Daniella Meeker, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-22-00479; P30AG024968 (NIH)
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Influenza; Vaccine Hesitancy
MeSH Terms: conditions — Influenza, Human; Vaccination Hesitancy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Texts (Active Comparator): Patients randomized to this study arm will receive a standard text reminding them about the importance of influenza vaccination. The standard texts will include a clinic call back number and patient portal self-scheduling for patients to schedule their influenza vaccines:
  #FirstName#, your flu shot is ready! Call your clinic at #ExternalRefNo# or visit the LA Health Portal at http://bit.ly/BookFluShot if you want this shot held for you.
  Interventions: Behavioral: Text messaging
- Standard Texts with Transportation messaging (Experimental): Patients randomized to this study arm will receive standard texts plus transportation messaging including a phone number for patients to reserve transportation to a vaccination appointment based on MediCal health plan transportation resources:
  #FirstName#, your flu shot is ready! Call your clinic at #ExternalRefNo# or visit the LA Health Portal at http://bit.ly/BookFluShot if you want this shot held for you. You can call #Health Plan Phone Number# to schedule a free ride for your flu shot through #HealthPlanName#.
  Interventions: Behavioral: Text messaging

INTERVENTIONS:
Behavioral: Text messaging — Patients will receive up to 3 text messages reminding them about the importance of influenza vaccination during the 2022-2023 flu season.

SUMMARY:
Previous studies have shown that low-cost, behavioral nudges through texting can increase influenza vaccination uptake compared to usual care. However, there are limited studies that evaluate the effect of decreasing barriers to scheduling, especially within safety net populations. The setting for this study, DHS, is the second largest public delivery system in the country and serves approximately half a million diverse patients that are eligible for vaccinations annually. This pilot study (one arm in a larger randomized controlled trial) will examine the effect of text messages highlighting MediCal health plan transportation resources (vs standard text messaging) on influenza vaccination rates in adults during the 2022-2023 flu season.

ELIGIBILITY:
Inclusion Criteria:

* Los Angeles County Department of Health Services (LACDHS) primary care patients over 6 months of age

Exclusion Criteria:

* LACDHS patients less than 6 months of age

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228831 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniella Meeker, PhD, Principal Investigator — University of Southern California
Locations (1):
- Los Angeles County Department of Health Services, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only one household member (index person) is randomized and all other members receive the same message
Groups:
- Standard Texts: Patients randomized to this study arm will receive a standard text reminding them about the importance of influenza vaccination. The standard texts will include a clinic call back number and patient portal self-scheduling for patients to schedule their influenza vaccines:
  #FirstName#, your flu shot is ready! Call your clinic at #ExternalRefNo# or visit the LA Health Portal at http://bit.ly/BookFluShot if you want this shot held for you.
  Text messaging: Patients will receive up to 3 text messages reminding them about the importance of influenza vaccination during the 2022-2023 flu season.
- Standard Texts With Transportation Messaging: Patients randomized to this study arm will receive standard texts plus transportation messaging including a phone number for patients to reserve transportation to a vaccination appointment based on MediCal health plan transportation resources:
  #FirstName#, your flu shot is ready! Call your clinic at #ExternalRefNo# or visit the LA Health Portal at http://bit.ly/BookFluShot if you want this shot held for you. You can call #Health Plan Phone Number# to schedule a free ride for your flu shot through #HealthPlanName#.
  Text messaging: Patients will receive up to 3 text messages reminding them about the importance of influenza vaccination during the 2022-2023 flu season.
Period: Overall Study
Arm/Group | Standard Texts | Standard Texts With Transportation Messaging
Started | 224959 | 3872
Completed | 224959 | 3872
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of the initial number randomized, only 124,793 had insurance that provided transportation benefits, and were therefore eligible for the transportation intervention and included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Texts | Standard Texts With Transportation Messaging | Total
Number analyzed (Participants) | 121743 | 3050 | 124793
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.27 (19.68) | 45.25 (19.78) | 45.27 (19.68)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 62819 | 1595 | 64414
  Sex/Gender: Male | 55271 | 1363 | 56634
  Sex/Gender: Unknown/Not reported | 3653 | 92 | 3745
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 69637 | 1741 | 71378
  Not Hispanic or Latino | 32141 | 776 | 32917
  Unknown or Not Reported | 19965 | 533 | 20498
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 121743 | 3050 | 124793

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Vaccinated at the End of the Campaign Period
Description: Number of Participants who received their influenza vaccination during the campaign period, as measured in the California Immunization Registry (CAIR2) to include vaccinations occurring both inside and outside the LADHS system. We assessed baseline vaccination status at the beginning of the flu season and excluded individuals who already received their vaccination.
Time Frame: 6 months
Population: As not all randomized participants were eligible for the transportation messaging given their insurance did not cover healthcare transportation costs, these households were removed from both groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Texts | Standard Texts With Transportation Messaging
Number analyzed (Participants) | 121743 | 3050
Participants | 33357 | 854
Statistical Analysis 1: Comparison: Standard Texts; Test type: Superiority; p = 0.216, 2 proportion Z-test; Percent Difference = .64

2. Secondary Outcome: Heterogeneity of Treatment Effects for Demographics
Description: Heterogeneity of treatment effects for demographic groups (previous vaccination status: vaccinated or unvaccinated)
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Texts | Standard Texts With Transportation Messaging
Number analyzed (Participants) | 121743 | 3050
Participants
  Previously vaccinated | 44742 | 1129
  Previously unvaccinated | 77001 | 1921
Statistical Analysis 1: Comparison: Standard Texts; Previously vaccinated; Test type: Superiority; p = 0.34, 2 proportion Z-test; Percent Difference = -0.61
Statistical Analysis 2: Comparison: Standard Texts; Previously unvaccinated; Test type: Superiority; p = 0.247, 2 proportion Z-test; Percent Difference = -0.45

ADVERSE EVENTS:
Time Frame: 6 months following messaging intervention
Description: Of the initial number randomized, only 124,793 (121,743 in Standard Text, and 3050 in Standard Text + Transportation) had insurance that provided transportation benefits, and were therefore eligible for the transportation intervention and included in the baseline analysis population. Therefore, we use these numbers when determining our At Risk population.
Arm/Group | Standard Texts | Standard Texts With Transportation Messaging
All-Cause Mortality (participants affected / at risk) | 0/121743 | 0/3050
Serious Adverse Events (participants affected / at risk) | 0/121743 | 0/3050
Other Adverse Events (participants affected / at risk) | 0/121743 | 0/3050

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT05537441/Prot_SAP_000.pdf